CLINICAL TRIAL: NCT02048033
Title: Medico-economic Evaluation of the Management of Weight Regain After Gastric Bypass by Gastrointestinal Narrowing of Jejunal Anastomosis by Endoscopic Suturing: Apollo Endosurgery OverStitch Technical
Brief Title: Assessment of the Overstich Technique for the Management of Weight Regain After Gastric Bypass.
Acronym: APOLLO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Following the occurrence of four serious adverse events in the APOLLO group and after discussion with the investigator, we consider that this minimally invasive protocol causes an increased risk of morbidity and mortality.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50372
Record Dates: First submitted 2014-01-16; First posted 2014-01-29 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: the Management of Weight Regain After Gastric Bypass by Endoscopic Suturing
Keywords: Obesity; Endogastric suturing; Jujenal anastomosis; weight regain
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm with Apollo Endosurgery OverStitch technical (Active Comparator)
  Interventions: Device: Regular endoscopy + endogastric suturing
- Arm without Apollo Endosurgery OverStitch technical (Placebo Comparator)
  Interventions: Diagnostic Test: Regular endoscopy

INTERVENTIONS:
Device: Regular endoscopy + endogastric suturing — Patients will get the usual endoscopy used for diagnosis. In addition, they will receive an endoscopic surgery using the APOLLO Endosuregery technique. The Apollo Endosurgery OverStitch is an endoscopic equipment which involves the suturing by endogastric way to decrease the size of the anastomosis gastrojujenal or gastric pouch
  Arms: Arm with Apollo Endosurgery OverStitch technical
Diagnostic Test: Regular endoscopy — Patients will get the usual endoscopy used for diagnosis.
  Arms: Arm without Apollo Endosurgery OverStitch technical

SUMMARY:
Prospective multicenters randomized study to compare the efficiency and the socioeconomic impact of the endoscopic management (Overstitch technique) of weight regain after gastric bypass surgery to non invasive treatment

DETAILED DESCRIPTION:
Nowadays morbid obesity (BMI ≥ 40kg/m²) is a major problem of public health in industrialized countries. About 500 000 patients would be affected by this disease in France in 2009. Prevalence of the morbid obesity raised from 0.3 % (± 0.1 %) of the population in 1997 to 1.1 % (± 0.1 %) in 2009 (Extrapolation of the data ObEpi on 2009 to the French population) (1). For this type of patient, the only long-term effective treatment recognized by the scientists is the bariatric surgery. (2-4) Roux and Y Gastric Bypass (GBP) is a consensual procedure, that has been described in the sixties, in this indication (approximately 11000 GBP performed in FRance in 2012 (5,6). This operation consists on the creation of a proximal gastric pouch (50 cc). A Roux and Y intestinal loop will be added to create a malabsorptive part. 60 to 80 % of excess weight loss described in the literature in the long-terms. Furthermore, improvement or remission of T2DM, sleep apnea syndrome, arterial hyperpressure, dyslipidemia) are emphasized in many trials (5, 7). However 15 to 20 % of the handled patients present a weight regain 5 years post surgery potentially explained by the dilation of the gastric pouch or the gastro jejunal anastomosis and thus a decrease of the restrictive effect. (8-11) To palliate this complication two solutions are described. (12-15; 19) The first one consists in a recalibration of the gastric poouch by surgical approachy. In this case, a ring of silicone or polypropylene can be positioned around the gastric pocket. Other possible solution is to redo a new gastrojejunostomy with a smaller size, by surgical access (laparotomy or laparoscopy). These interventions are very delicate because of important peritoneal adhesions and present a rate of significant morbidity especially if they are performed under laparotomy. The pure medical care does not allow long-term results stable. ²² A therapeutic dead end is reported often for this type of patient. A new possibility was recently described. (17-18) A recalibration can be realized by sutures performed under endoscopic approach at the level of the gastro jejunal anastomosis or from the gastric pouch by the APOLLO Endosurgery OverStitch. The digestive surgery by endoscopic way is rapidly expanding. The first results seem to be promising (resumed the weight loss) but owe to be estimated in a randomized study comparing this new process with the medical conventional treatment. A single-blind, randomized, forward-looking study, multicenter, comparative between two parallel groups of patients presenting a weight regain after GBP was thus organized. The main objective is to estimate the efficiency of the APOLLO Endosurgery OverStitch technique versus the non-interventional strategy. The secondary endpoints is to study the morbidity of the procedure, the evolution of quality of life of the patients, the medical economic impact of the innovation in 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Surgical criteria: patient with bariatric surgery by gastric bypass since, at least, 24 months
* Clinics criteria of weight regain or treatment failure:

  * Patient with weight regain> 5kg / m²
  * Patient with EWL (excess weight loss) <25% after 2 years of treatment.
* Loss of early satiety (interrogation)
* Patient with a compatible psychological and cognitive status with the study,
* Patient agreeing to follow the procedures of the study and can participate at the follow-up study during 2 years
* Subject with no rights from the national health insurance programme
* Consent form signed

Exclusion criteria:

* Pregnancy (plasma assay of beta-HCG positive)
* Presence of cardiovascular, neurological, psychiatric, endocrine, renal, gastrointestinal or tumor comorbidities making irrelevant patient participation in the judgment of the investigator
* Patient participating in another clinical study or participated in another study within the last 30 days or for which the annual compensation received exceeds € 4,500
* Patient with a contre-indication to the achievement of surgery (fistula, ulceration, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Weight loss assessment of Apollo Endosurgery OverStitch technical | At 12 and 24 months after surgery
  The main objective is to compare the efficacy of endoscopic surgery Apollo Endosurgery OverStitch technical than the conventional non-interventional strategy in patients with weight regain after gastric bypass.Moreover, all of these patients will also benefit from the medical-nutritional usual care.

SECONDARY OUTCOMES:
Comparison of both strategies on tolerance (adverse events and serious adverse events) | At 12 months after Baseline and at each visit
  The secondary objectives of this study were to compare in real life these both strategies of the management of weight regain after gastric bypass on tolerance and safety related to obesity.
Comparison of both strategies on comorbidities | At 12 months after Baseline and at each visit
  The secondary objectives of this study were to compare in real life these both strategies of the management of weight regain after gastric bypass on comorbidities related to obesity (type 2 diabetes, arterial hypertension, sleep apnea syndrome, ...).
Comparison of both strategies on quality of life | At 12 months after Baseline and at each visit
  The secondary objectives of this study were to compare in real life these both strategies of the management of weight regain after gastric bypass on quality of life.
Comparison of both strategies on medico-economic impact (drugs fees, medical consultation fees..) | At 12 months after Baseline and at each visit
  The secondary objectives of this study were to compare in real life these both strategies of the management of weight regain after gastric bypass on medico-economic impact of innovation.
  Moreover, a cost-effectiveness analysis will be performed at the end of this study.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Louis Mourier Hospital, Colombes
  - Lille Hospital, Lille
  - Montpellier Hospital, Montpellier
  - Nice Hospital, Nice
  - HEGP Hospital, Paris
  - Strasbourg Hospital, Strasbourg
  - Villeurbanne clinic, Villeurbanne